CLINICAL TRIAL: NCT00572650
Title: An Open-label, Parallel-group Study to Determine the Single and Multiple Dose Pharmacokinetics of LAF237 and Its Metabolites in Mild Renal Impaired Patients Compared to Age, Sex and Weight-matched Healthy Volunteers Following Daily Doses of 100 mg LAF237 for 14 Days
Brief Title: Pharmacokinetic Study of LAF237 and Its Metabolites in Mild Renal Impaired Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237A2117
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type-2 diabetes, DPP-4 inhibitor, vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator)
  Interventions: Drug: vildagliptin

INTERVENTIONS:
Drug: vildagliptin — 16 volunteers in each group of mild renal impairment patients and their matched healthy volunteers will receive once daily doses of 100mg LAF237 for 14 days.

SUMMARY:
This study will evaluate the pharmacokinetics of vildagliptin (LAF237) and its metabolites in patients with mild renal impairment compared to their sex, age and weigh based healthy volunteer counterparts.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years of age (inclusive).
* Male, non-fertile female or female of childbearing potential using a medically approved birth control method.
* Body mass index (BMI) ≤42 kg/m2 (inclusive) at Screening.
* Able to provide written informed consent prior to study participation.
* Able to communicate well with the investigator and comply with the requirements of the study.

For renal insufficient patients only

* Patients must have stable renal disease without evidence of renal progressive disease
* If patient is diabetic, must be treated with standard anti-diabetic therapy andmust agree to continue their anti-diabetic therapy throughout the duration of the study.
* If patient is diabetic, must be on a stable dose of standard anti-diabetic therapy or diet and exercise regimen over the past 4 weeks prior to Screening.

For healthy subjects only

* No current significant medical conditions as determined by history and physical.
* A serum creatinine with a calculated CrCl of >80 ml/min.
* Matched to renal impaired patients (Group A) undergoing study by age (±5 years), sex and weight (±10% BMI).

Exclusion Criteria:

Subjects meeting any of the following criteria during screening or baseline evaluations will be excluded from entry into or continuation in the study:

* Pregnant or lactating female.
* A history of certain disorders as specified in the protocol.
* Subjects that have been enrolled in a LAF237 (vildagliptin) study or other DPP-4 inhibitor studies six months prior to Baseline.
* History of renal transplant at any time in the past and on immunosuppressant therapy.
* Acute infections which may affect blood glucose control within 4 weeks prior to Screening and other concurrent medical condition that may interfere with the interpretation of efficacy and safety data during the study.
* Certain electrocardiogram (ECG) abnormalities:
* Malignancy including leukemia and lymphoma (not including basal cell skin cancer) within the last 5 years.
* Liver disease such as cirrhosis or positive hepatitis B and C.
* Any alcohol related hepatic disease.
* Patients undergoing any method of dialysis (hemodialysis or peritoneal dialysis)
* Concurrent medical condition that may interfere with the interpretation of safety and tolerability data during the study.
* Use of certain medications as specified in the protocol.
* Laboratory abnormalities as defined by the protocol
* History of active substance abuse (including alcohol) within the past 2 years.
* Smokers defined as any subject who reports heavy cigarette use (i.e., 10 or more cigarettes per day). Urine cotinine will also be measured and recorded at Screening and Baseline.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic measures | throughout the study

SECONDARY OUTCOMES:
Safety and tolerability measures | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: NOVARTIS, Principal Investigator — Novartis investigator site
Locations (1):
- Novartis Investigator Site, Kiel, Germany